CLINICAL TRIAL: NCT05086341
Title: A Randomized Controlled Pilot- and Feasibility Trial of the EHealth Tool My COPD, to Evaluate User Satisfaction, Reach and Safety in People with Chronic Obstructive Pulmonary Disease
Brief Title: A Pilot- and Feasibility Trial of the EHealth Tool My COPD for People with COPD
Acronym: My COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Feasibility My COPD; 2020-01957 (Other Grant/Funding Number: The Swedish Research Council); 20190406 (Other Grant/Funding Number: The Swedish Heart and Lung Foundation); RV-939255 (Other Grant/Funding Number: Alf-Grant Region Västerbotten)
Record Dates: First submitted 2021-09-26; First posted 2021-10-20 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2023-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Telemedicine; Telerehabilitation; eHealth; Participatory; Exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Intervention Model Description: Parallel-group, randomized controlled pilot- and feasibility trial, 2:1 (I:C) randomization.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- My COPD (Experimental): In addition to usual care, participants in the intervention group will receive a 12-week, twice a week, physiotherapist-supported individualized exercise program and physical activity plan via the eHealth tool My COPD.
  Interventions: Device: My COPD
- Usual care (No Intervention): Participants in the control group will receive usual care only. Usual care is recommended to include, but not restricted to, long-acting anticholinergics and long-acting ß2-antagonists with 24-hour duration and support for smoking cessation, PA and exercise, self-management and nutrition.

INTERVENTIONS:
Device: My COPD — In addition to usual care, participants in the intervention group will initially meet with a physiotherapist to set up an individualized exercise program and physical activity plan. Participants will also receive a device instruction manual and a one hour of face-to-face training on how to use My COPD. The 12-week intervention is home-based, and self-managed with support from physiotherapist via My COPD. In addition to warm-up exercises, the exercise program comprises five exercises targeting major muscle groups, as well as, balance and aerobic exercise, to be conducted at least twice weekly. Via My COPD, the physiotherapists can follow activities and progress the exercise program, and the physiotherapist and the participants can contact each other. Throughout the intervention period, technical support will be available.
  Arms: My COPD

SUMMARY:
The aim of this multi-center, randomized controlled pilot- and feasibility trial is to evaluate the user satisfaction, reach and safety of My COPD, a novel eHealth tool for remote delivery of evidence-based treatment targeting people with chronic obstructive pulmonary disease (COPD). In addition, the investigators aim to collect and synthesize data on clinical outcome measures to inform the sample size estimation of a later, definitive trial.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is one of the most common non-communicable (chronic) diseases, leading to significant increased risk of morbidity and mortality. Pulmonary rehabilitation is a comprehensive intervention, including but not limited to physical exercise, education and behavioral change. Conclusive evidence supports the provision of pulmonary rehabilitation in adults with COPD, which benefits exercise tolerance, physical activity, health-related quality of life, health care use, and survival. However, access to pulmonary rehabilitation needs to be increased, which has recently been highlighted as a top priority by leading experts in the area.

To increase access to evidence-based treatment for people with COPD this research group has developed a novel eHealth tool, My COPD, in co-creation with intended end-users to meet requirements and needs of adults with COPD and health care providers. My COPD includes components to promote physical exercise, education and behavioral change, for example, information on disease management and treatment, symptom diary, an individualized physical exercise and activity plan, support from physiotherapist as well as self-management strategies. My COPD will be available on a nation-wide platform for internet-based support- and treatment programs that regional health care regions throughout Sweden offers.

The research aim of this trial is to explore the users' satisfaction, reach and safety of My COPD, and to collect and synthesize data on clinical outcome measures to inform the sample size estimation of a later definitive trial. For this purpose, the investigators will conduct a multi-center, parallel-group randomized controlled pilot- and feasibility trial, with usual care as comparison group (control), for the duration of 12 weeks. In total, 30 adults with stable COPD will be recruited from hospitals and primary care centers located in public health regions in central (Region Stockholm) and northern (Region Västerbotten) Sweden.

All participants will be invited to complete an initial screening and baseline assessment before the randomization and intervention commences. Descriptive baseline assessments that will be collected include assessment of pulmonary function (spirometry), while having usual bronchodilator therapy according to guidelines. Anthropometric data collected will include age, sex, height, weight, and body mass index. Further data that will be collected include information on smoking status, education, and co-morbidities and medications that may influence physical capacity or activity.

At completion of informed consent, enrolment and baseline assessment procedures, participants will be randomized to either the intervention group (My COPD) or control group (usual care). Randomization will be conducted using opaque envelopes, and administered by a researcher not involved in the assessment procedures, thus, ensuring concealed allocation. Participants will be randomized to the intervention (My COPD) and control group (usual care) group, using a 2:1 allocation ratio and stratified by sex and center.

Before and after the 12-week intervention assessments of exercise capacity, balance, level of physical activity, health related quality of life, COPD related symptoms, health economics will be conducted in all participants. During the intervention, data on exercise intensity, adverse events, adherence and progression will be collected from participants in the intervention group via My COPD. At intervention completion the user satisfaction of participants and health care professionals in the intervention group will be assessed. Participants in both groups will be asked to describe their COPD-related health care contacts during the study period. Physiotherapists, blinded to group allocation and previous test results, will conduct assessments.

ELIGIBILITY:
Inclusion Criteria:

* a confirmed diagnosis of COPD

Exclusion Criteria:

* inability to read and understand Swedish
* severe comorbidity that can be considered as the main contributing factor for limitation in physical activity.

In case of an exacerbation, the participant has to wait six weeks from the start of pharmacological treatment before being eligible in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
User satisfaction | 12-week follow-up (end of intervention)
  The mHealth App Usability Questionnaire (MAUQ) for patients, and health care staff, with score ranging 21-147 (higher score indicating better usability)

SECONDARY OUTCOMES:
Physical capacity | Baseline and 12-week follow-up
  The 6 minute walk test (6MWT) (distance in meters)
Physical capacity | Baseline and 12-week follow-up
  The 1 minute sit-to-stand test (count)
Physical capacity | Baseline and 12-week follow-up
  The Timed Up and Go (TUG) (time in minutes)
Physical capacity | Baseline and 12-week follow-up
  The Unsupported Upper Limb Exercise test (UULEX)(time in minutes)
Level of physical activity | Accelerometer wear (7 days prior to intervention commencement) and at 12-week follow-up
  Accelerometer (Minimod, McRoberts®, NL) (steps, time in activity/inactivity)
Level of physical activity | Baseline and 12-week follow-up
  Indicator questions on physical activity (time in hours)
Health related quality of life (HrQoL) | Baseline and 12-week follow-up
  The St Georges Respiratory Questionnaire (SGRQ), with score ranging from 0-100 (higher score indicating more limitation)
COPD related symptoms | Baseline and 12-week follow-up.
  The Modified Medical Research Council dyspnea scale (mMRC), with score ranging 0-4 (higher score indicating more symptoms)
COPD related symptoms | Baseline and 12-week follow-up.
  The COPD Assessment test (CAT), with score ranging 0-40 (higher score indicating more symptoms)
Health economics | Baseline and 12-week follow-up
  The EQ-5D to estimate change in quality-adjusted-life-years (QALYs), with score ranging 0-100 (higher score indicating better health)
Health economics | During the 12-week intervention
  Frequency of self-reported COPD-related health care contacts to estimate health care use (counts)

OTHER OUTCOMES:
Exercise intensity | During the 12-week intervention
  The Borg CR-10, with a score ranging 0-10 (higher score indicating higher intensity)
Adverse events | During the 12-week intervention
  Frequency and severity
Adherence | During the 12-week intervention
  Frequency of completed exercise sessions/activities
Progression of exercises | During the 12-week intervention
  Frequency of completed exercise levels

CONTACTS AND LOCATIONS:
Overall Officials: Karin Wadell, PhD, Principal Investigator — Umeå University
Locations (2):
- Sweden (2):
  - Karolinska Intitutet, Stockholm
  - Umeå university, Umeå

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karlsson A, Sonnerfors P, Lundell S, Toots A, Wadell K. Evaluation of a Novel eHealth Tool for Pulmonary Rehabilitation in People With Chronic Obstructive Pulmonary Disease: Randomized Controlled Pilot and Feasibility Trial. JMIR Form Res. 2025 Jun 23;9:e68195. doi: 10.2196/68195. PMID 40550122